CLINICAL TRIAL: NCT05100264
Title: Effect of Acidic Vaginal pH on the Efficacy of Dinoprostone (PGE2) Vaginal Tablet for Labor Induction in Full Term Pregnant Women: A Randomized Controlled Trial
Brief Title: Effect of Acidic Vaginal pH on the Efficacy of Dinoprostone for Labor Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandra Hospital, Athens, Greece (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Georgios Daskalakis, Professor of Obstetrics and Gynecology, Alexandra Hospital, Athens, Greece
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 68/7/22-9-21
Record Dates: First submitted 2021-10-18; First posted 2021-10-29 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Labor, Induced; Induced; Birth
Keywords: labor induction; dinoprostone; vaginal pH
MeSH Terms: interventions — Acetic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be computer generated. Allocation concealment will be ensured by opaque sealed envelopes. Blinding of outcomes assessor, principal as well as other investigators will be ensured as randomization will be performed by an external investigator that will not participate in the clinical process of the study or the statistical analysis. The ward midwife will open the randomization envelope after patient enrollment and different types of vaginal washing will be applied as per randomization. Participant as well outcomes assessor (physician that will evaluate the progress of labor as well statistician involved in the analysis) will be blinded to the procedure.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal washing 5% acetic acid (Experimental)
  Interventions: Other: Vaginal washing with 5% acetic acid
- Vaginal washing 0.9% N/S (Placebo Comparator)
  Interventions: Other: Vaginal washing with 0.9% NS

INTERVENTIONS:
Other: Vaginal washing with 5% acetic acid — Induction of labor (vaginal tablet dinoprostone and vaginal washing with 5% acetic acid)
  Arms: Vaginal washing 5% acetic acid
Other: Vaginal washing with 0.9% NS — Induction of labor (vaginal tablet dinoprostone and vaginal washing 0.9% NS)
  Arms: Vaginal washing 0.9% N/S

SUMMARY:
Acidification of vaginal pH has been proposed as a potential factor that could help increase the efficacy of vaginal prostaglandins in labor induction. The aim of the present randomized controlled trial is to evaluate the impact of an acidic vaginal pH on the progress of labor induction with dinoprostone (Prostaglandin E2 - PGE2) vaginal tablet.

ELIGIBILITY:
Inclusion criteria

* Singleton pregnancy
* Full term (>37 weeks)
* Cephalic presentation
* Reactive NST (nonstress test)
* Absence of spontaneous uterine contractions
* No contraindications to vaginal delivery

Exclusion criteria

* Multifetal pregnancy
* Fetal malpresentation
* Preterm delivery (<37 weeks)
* Advanced maternal age (>40 years)
* Bishop score > 7
* Fetal macrosomia ( >4500 gr)
* Non reassuring NST (nonstress test)
* Suspected chorioamnionitis
* Previous cesarean delivery or other uterine surgery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 230 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Interval from induction to delivery | 36 hours
  Time interval (minutes)

SECONDARY OUTCOMES:
Interval from induction to active labor | 36 hours
  Time interval (minutes)
Interval from induction to second stage of labor | 36 hours
  Time interval (minutes)
Failure of induction of labor | 36 hours
  Rate of participants with failure of induction of labor

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Daskalakis, Study Director — Alexandra General Hospital
Locations (1):
- Alexandra General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided